CLINICAL TRIAL: NCT04566536
Title: NoL Monitor Performances of Nociceptive and Non-nociceptive Stimuli Discrimination During Robotic Surgery Under Propofol-remifentanil Anaesthesia
Brief Title: NoL Monitor Performances of Nociceptive and Non-nociceptive Stimuli Discrimination During Robotic Surgery
Acronym: ROBOTNOL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191091; 2019-A02744-53 (Other: IDRCB)
Record Dates: First submitted 2020-09-14; First posted 2020-09-28 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Pain Management
Keywords: NoL; Nociception; Robotic surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: Patients ≥ 18 years old scheduled for robotic surgery (all specialties except ENT)

SUMMARY:
Anesthesia quality and safety have improved over the past decades, thanks to improved monitoring devices. No nociception monitoring is currently part of the standard of care. Usually, hemodynamic parameters are used to evaluate nociception (heart rate, HR, and mean arterial pressure, MAP), but none of them are specific. However, nociception evaluation is critical. Indeed, where excess of nociception can lead to arterial hypotension and respiratory depression, insufficient nociception can lead to acute postoperative pain, which is followed by persistent chronic pain in 10-50% of patients. Different monitoring devices have been developed but none of them are still used in current practice. Recently developed, the nociception level (NoL) index (MEDASENSE BIOMETRICS Ltd®, Ramat Gan, Israel) is an index of nociception, based on a nonlinear algorithm combination of heart rate, heart rate variability, photoplethysmograph wave amplitude, skin conductance, skin conductance fluctuations, and their time derivatives.

Robotic surgeries have started to spread over the world 20 years ago, claiming to be mini-invasive with less hemorrhage complications, with better success based on the technical advantages of the robot allowing better access during anatomical challenges procedures. Robotic surgery has been suggested to decrease pain during surgery and post-operatively, because of the decreases abdominal wall constraints induced by the robotic arms compared to the surgeon arms.

This observational prospective non-interventional monocentric study intend to evaluate the performance of the NoL index to discriminate protocol-defined nociceptive from non nociceptive stimuli during robotic surgery.

All patients, scheduled for a robotic surgery procedure, will be orally informed about the study during the anesthesia consultation. During the procedure, the anesthesia procedure will be the same for all patients, as part of the usual care in our department. The NoL monitor will be added for the purpose of this study, but the results will be hidden from all physicians. All settings will be left the physician in charge. At the end of the surgical procedure, before transfer to the recovery room, data for the monitor will be extracted on a dedicated universal serial bus (USB) key. Files will be safely stored under RedCap before analysis.

DETAILED DESCRIPTION:
Anesthesia quality and safety have improved over the past decades, thanks to improved monitoring devices. Excess of anesthetics could lead to arterial hypotension which has been shown to be associated with increased cardiovascular events. On the other hand, insufficient anesthetics could lead to awareness and memorization during general anesthesia (GA). Whereas almost all drugs currently used in the operating room (OR), have a validated monitoring tool, no nociception monitoring is currently part of the standard of care. Usually, hemodynamic parameters are used to evaluate nociception (heart rate (HR), and mean arterial pressure (MAP)), but none of them are specific and several factors in the OR influence these parameters. There is growing interest in the literature for nociception monitoring. Indeed, where excess of nociception can lead to arterial hypotension and respiratory depression, insufficient nociception can lead to acute postoperative pain, which is followed by persistent chronic pain in 10-50% of patients. Opioids per se can also induce nausea and vomiting, hyperalgesia for remifentanil.

Different monitoring devices, like the surgical pleth index, pupillometry or the "Analgesia Nociception Index", have been developed, based on several variables and algorithms, but none of them are still used in current practice. One of the major reason is that although they might had some effects on clinical parameters or drugs consumption, none of them had any influence on patient outcome. Recently developed, the nociception level (NoL) index (MEDASENSE BIOMETRICS Ltd®, Ramat Gan, Israel) is an index of nociception, based on a nonlinear algorithm combination of heart rate, heart rate variability, photoplethysmograph wave amplitude, skin conductance, skin conductance fluctuations, and their time derivatives. One of the first study to report the ability of the NoL index to discriminate noxious from non-noxious stimuli with high sensitivity and specificity was performed in 2016. In that randomized trial (continuous infusion of remifentanil target 2 versus 4 ng/ml) enrolling 58 patients undergoing a large range of surgery, the NoL index was superior than the hemodynamic parameters alone to characterize nociception. In a study enrolling 72 patients randomized within 6 remifentanil concentration targets undergoing several surgical procedures by the same authors, the NoL index was not affected by remifentanil doses, whereas it had an dose-dependent hemodynamic effect on HR and MAP.

Robotic surgeries have started to spread over the world 20 years ago, claiming to be mini-invasive with less hemorrhage complications, with better success based on the technical advantages of the robot allowing better access during anatomical challenges procedures. Debates recently arise based on the procedures cost and the little (or lack) of evidence of mini-invasive procedures in patients with cancers. Robotic surgery has been suggested to decrease pain during surgery and post-operatively, in gynecologic, thoracic, and general procedures although results are controversial, because of the decreases abdominal wall constraints induced by the robotic arms compared to the surgeon arms. To our knowledge, none of these studies evaluated pain based on a nociception monitoring device.

This observational prospective non-interventional monocentric study intend to evaluate the performance of the NoL index to discriminate nociceptive from non nociceptive stimuli during robotic surgery.

All patients, scheduled for a robotic surgery procedure, will be orally informed about the study during the anesthesia consultation. During the procedure, the anesthesia procedure will be the same for all patients, as part of the usual care in our department. Patients will be closely monitored by electrocardiogram, intermittent blood pressure by arm cuff, continuous pulse oximetry by finger probe, neuromuscular monitoring by train-of-four (TOF)-Cuff, bispectral index (BIS) monitoring using the BIS forehead 4-sensor. The NoL monitor will be added for the purpose of this study, but the results will be hidden. The probe will be placed on the hand contralateral to the blood pressure arm cuff. Anesthesia will be delivered by target-controlled infusion of remifentanil and propofol by two separate infusion pumps. Once consciousness will be lost and a TOF calibration done, neuromuscular blockade will be performed by rocuronium 0.6 mg/kg. All settings will be left the physician appreciation. Different stimuli (nociceptive and non-nociceptive) are defined according to protocol (such as intubation, incision, surgical haemostasia, urinary track catheter…) and their time of arrival will be collected in a Case Report Form. At the end of the surgical procedure, before transfer to the recovery room, data for the monitor will be extracted on a dedicated USB key. Files will be safely stored under RedCap before analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Scheduled for a robotic surgery in the center of investigation (all specialties except cardiac and ENT: gynaecologic, thoracic, urologic and abdominal)
* Non-opposition to the study participation

Exclusion criteria :

* Age < 18 years old
* Rapid sequence anaesthesia required
* Pregnancy and breast feeding
* Chronic medication by any pain killer (opioids or not)
* ENT and cardiac robotic surgery
* Neuromuscular disease
* NoL Index contre-indications, such as cardiac arrythmia, supra-clavicular arterial stenosis, severe hypovolemia, severe hypothermia
* Chronic alcoholism, toxicomania
* Severe obesity (IMC > 35)
* Legal protection
* Opposition to the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robotic surgery in Bichat Hospital, APHP, Paris, France
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
NoL index validation | 7 hours
  Area under the curve with the 95% confidence interval, based on the NoL absolute value after nociceptive and non-nociceptive stimuli.

SECONDARY OUTCOMES:
Discriminative diagnosis performance (nociceptive from non-nociceptive stimuli) of the heart rate after nociceptive and non-nociceptive stimuli. | 7 hours
  Sensitivity, specificity and area under the curve
Discriminative diagnosis performance (nociceptive from non-nociceptive stimuli) of the mean arterial pressure | 7 hours
  Sensitivity, specificity and area under the curve of the mean arterial pressure after nociceptive and non-nociceptive stimuli.
Discriminative diagnosis performance (nociceptive from non-nociceptive stimuli) of the BIS index | 7 hours
  Sensitivity, specificity and area under the curve of the BIS index after nociceptive and non-nociceptive stimuli.
Correlation between the NoL index and the mean arterial pressure during nociceptive stimuli | 7 hours
  Spearman correlation test within the NoL index variations and the mean arterial pressure variations after each stimuli
Correlation between the NoL index and the heart rate during nociceptive stimuli | 7 hours
  Spearman correlation test within the NoL index variations and the heart rate variations after each stimuli
Delay of the NoL index to detect a nociceptive stimuli | 7 hours
  Delay between a NoL index above 25 and the nociceptive stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie GOUEL-CHERON, MD, PhD, Principal Investigator — Hôpital Bichat-Claude Bernard, AP-HP
Locations (1):
- Hôpital Bichat-Claude Bernard, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No